CLINICAL TRIAL: NCT01460849
Title: Assess the Increased Mortality Risk With Each Year of Delayed TIS Initiation, and the Effect of TIS on Mortality Across Study Centers
Brief Title: Assess Increased Mortality Risk With Each Year of Delayed Tobramycin Solution (TIS) Initiation, and Effect of TIS on Mortality Across Study Centers
Status: Withdrawn | Type: Observational
Why Stopped: company decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: HEORUS0088
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Using CFF registry data, this analysis will: describe patterns of time to TIS initiation from first year of TIS eligibility, estimate the increased risk of death attributable to each year of delayed TIS initiation, and investigate TIS effects across study centers.

ELIGIBILITY:
Inclusion Criteria:

* ≥6 years of age with a documented Cystic fibrosis (CF) diagnosis,
* moderate-to-severe lung disease,
* Pseudomonas aeruginosa (PA) airway infection.

Exclusion Criteria:

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-03 (Estimated); Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Time to tobramycin solution (TIS) initiation from first year of TIS eligibility

SECONDARY OUTCOMES:
Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals